CLINICAL TRIAL: NCT03703414
Title: Characterization of Microbial, Immune and Epigenetic Biomarkers for Major Depressive Disorder and ECT Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0069-18-ZIV
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will obtain fecal samples and blood samples from participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Healthy controls
  Interventions: Diagnostic Test: Fecal microbiota composition analysis and blood cytokine level analysis
- ECT: MDD patients receiving ECT treatment
  Interventions: Diagnostic Test: Fecal microbiota composition analysis and blood cytokine level analysis
- SSRI: MDD patients receiving SSRI treatment
  Interventions: Diagnostic Test: Fecal microbiota composition analysis and blood cytokine level analysis

INTERVENTIONS:
Diagnostic Test: Fecal microbiota composition analysis and blood cytokine level analysis — Fecal microbiota composition analysis and blood cytokine level analysis

SUMMARY:
The investigators aim to characterize fecal microbial biomarkers as well as blood cytokine levels in MDD patients vs. healthy controls. 40 MDD patients will be recruited for this study, as well as 20 healthy age-matched participants (as a control group). Following signing of informed consent, stool and blood (20 ml) samples will be collected from all participants, for microbial composition assessment, and blood measures of inflammation and protein expression. According to clinical assessment of the diagnosed MDD patients, the psychiatrist will recommend SSRI or ECT treatment, and the patients will be divided accordingly to treatment group. Clinical status will be assessed by the Hamilton Depression Rating Scale (HAM-D) scored by a psychiatrist at the starting point (before treatment), after 4 weeks of treatment (as ECT-group patients receive 8-12 treatments on average). A lowering in the HAM-D score will be considered clinical improvement which may be attributed to treatment. The investigators expect a treatment success rate of over 50% for ECT according to past experience. Blood and stool samples will be collected from MDD patients after 4 weeks of treatment, repeating inflammatory, protein expression and microbial measurements and comparing them to initial results. Additional data recorded will include age, BMI, ethnicity, previous medication use, and number of ECT treatments or current medication.

DETAILED DESCRIPTION:
All procedures will be approved by the ZIV Helsinki ethics committee. Recruitment and clinical assessment: 40 MDD patients will be recruited for this study, as well as 20 healthy age-matched participants (as a control group). A psychiatrist not involved in the study will assess the qualification of the patients for signing informed consent. Following signing of informed consent, stool and blood (20 ml) samples will be collected from all participants, for microbial composition assessment, and blood measures of inflammation and protein expression. According to clinical assessment of the diagnosed MDD patients, the psychiatrist will recommend SSRI or ECT treatment, and the patients will be divided accordingly to treatment group. Clinical status will be assessed by the Hamilton Depression Rating Scale (HAM-D) scored by a psychiatrist at the starting point (before treatment), after 4 weeks of treatment (as ECT-group patients receive 8-12 treatments on average). A lowering in the HAM-D score will be considered clinical improvement which may be attributed to treatment. The investigators expect a treatment success rate of over 50% for ECT according to our past experience. The investigators will collect blood and stool samples from MDD patients after 4 weeks of treatment, repeat inflammatory, protein expression and microbial measurements and compare them to initial results. Additional data recorded will include age, BMI, ethnicity, previous medication use, and number of ECT treatments or current medication.

Inclusion criteria: MDD patients with stable depression clinically diagnosed by a psychiatrist according to the Hamilton Depression Scale. Patient age may range between 18-80 years, as depression is more common in older people as represented by a median age of over 55 in the treated population at the Ziv Medical Center.

Exclusion criteria: Patients receiving antibiotics in the past 3 months prior to sampling, patients suffering from chronic gastrointestinal diseases or other chronic diseases such as autoimmune or cancer, patients with comorbidities such as schizophrenia.

Blood samples: Whole blood will be centrifuged and serum samples will be kept at -80C until analysis for inflammatory measurements. Additionally, lymphocytes will be purified, RNA will be extracted and qRT-PCR will be performed to test immune protein and receptor expression (IL-1β, IL-1R1, IL-6, TNF-α, TNF1, TNF2) as well as additional proteins related to MDD (e.g. cannabinoid receptor 1- CNR1, CD38, oxytocin receptor- OXTR, brain-derived neurotrophic factor - BDNF).

Inflammatory measures in the serum: We will measure levels of pro and anti-inflammatory cytokines by multiplex tests including IL-1, IL-6, IL-8, IL-10, and TNFα using a Bio-Plex kit (Bio-Rad). The assay plate will be read on a MAGPIX multiplex reader (Bio-Rad).

Stool samples: stool samples will be stored within 4 hours from collection at -80C until processing.

Microbial analysis: Microbial DNA will be purified from stool and a barcoded 16S rRNA library from each subject will be generated from which we will obtain ~300,000 reads per sample using the Illumina MiSeq platform (NGS sequencing) at the Faculty of Medicine, Bar Ilan University. Sequences will be analyzed by QIIME. Additionally, microbial RNA will be extracted from stool in order to test microbial gene expression via metatranscriptomics (NGS sequencing).

Statistical analysis: All assays will be conducted using statistical software SPSS version 24 (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls
* MDD patients with stable depression clinically diagnosed by a psychiatrist according to the *Hamilton Depression Scale.
* Ages 18-80

Exclusion Criteria:

* Patients receiving antibiotics in the past 3 months prior to sampling
* Patients suffering from chronic gastrointestinal diseases
* Patients with chronic diseases such as autoimmune or cancer
* Patients with psychiatric co-morbidities such as schizophrenia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 MDD patients will be recruited for this study, as well as 20 healthy age-matched participants (as a control group).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between MDD and fecal microbial communities (as determined by NGS sequencing) and as well as immune components (cytokine levels in blood) | 4 week followup
Correlation between ECT treatment and fecal microbial communities (as determined by NGS) as well as blood cytokines in MDD patients | 4 week followup
Correlation between SSRI treatment and fecal microbial communities (as determined by NGS) as well as blood cytokines in MDD patients | 4 week followup

IPD SHARING:
Plan to Share IPD: No